CLINICAL TRIAL: NCT02344914
Title: Dental Support and the Second Stage of Labor Among Multiparous Women
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yariv yogev (Other)
Responsible Party: Sponsor-Investigator, Yariv yogev, Yariv Yogev, professor Director, division of obstetrics and delivery ward, Rabin Medical Center
Organization: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0523-14-RMC
Record Dates: First submitted 2014-12-21; First posted 2015-01-26 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-01

CONDITIONS: Second Stage of Labor
Keywords: dental support; second stage of labor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- receive Laboraide (Experimental): After giving consent, randomization will be carried out using sealed envelopes. After randomization women will be offered to withdraw consent. Women assigned to the study group will receive a sealed Laboraide™ package.
  Interventions: Device: receive Laboraide
- do not receive Laboraide (No Intervention): After giving consent, randomization will be carried out using sealed envelopes. After randomization women will be offered to withdraw consent. Women assigned to the control group.

INTERVENTIONS:
Device: receive Laboraide — After giving consent, randomization will be carried out using sealed envelopes. After randomization women will be offered to withdraw consent. Women assigned to the study group will receive a sealed Laboraide™ package.
  Labor follow up will be documented regularly including outcome. The use of the DSD will not affect the regular management of labor according to the routine standards of the delivery suite. Following delivery, patients will be asked to complete a satisfaction questionnaire.
  Arms: receive Laboraide

SUMMARY:
To assess if the use of the dental support device( DSD) Laboraide™ shortens the second stage of labor and decreased the rate of obstetrical interventions, and if it's use alleviate pain.

DETAILED DESCRIPTION:
Several studies have demonstrated that a dental support device (DSD) may increase the isometric strength of different muscle groups (1-7). A preliminary pilot study of 32 women in 2009 showed that DSD may shorten the second stage of labor among nulliparous women (8) by increasing the expulsive efforts of the parturient. The study hypothesis was that DSD may decrease the length of the second stage of labor and decrease the need for obstetrical interventions such as cesarean delivery or operative vaginal delivery.

The Laboraide™ is a DSD developed specifically for use during labor. It is an inert device located between the jaws and does not interfere with speaking, breathing or any other oral activity during labor. It is a single use device, and is not transferred between women. We hypothesize that using this device can shorten the second stage of labor and decrease obstetrical intervention rate. We will also investigate it's efficiency in pain management.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton gestation
2. Multiparous women
3. Term gestation (>37+0/7 weeks)
4. Signed written consent to participate in the study
5. Maternal age 18-45 years
6. Normal vital signs
7. Noraml cardiotocography and biophysical profile at admission

Exclusion Criteria:

1. Multiple gestation
2. Nulliparous women
3. preterm gestation (<37+0/7 weeks)
4. Refusal to participate
5. Maternal age <18 or > 45 years
6. Normal vital signs
7. Abnormal cardiotocography and biophysical profile at admission

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Duration of the second stage of labor. | 12 month
  After giving consent, randomization will be carried out using sealed envelopes. After randomization women will be offered to withdraw consent. Women assigned to the study group will receive a sealed Laboraide™ package.
  Labor follow up will be documented regularly including outcome. The use of the DSD will not affect the regular management of labor according to the routine standards of the delivery suite. Following delivery, patients will be asked to complete a satisfaction questionnaire.
Mode of delivery. | 12 month
  After giving consent, randomization will be carried out using sealed envelopes. After randomization women will be offered to withdraw consent. Women assigned to the study group will receive a sealed Laboraide™ package.
  Labor follow up will be documented regularly including outcome. The use of the DSD will not affect the regular management of labor according to the routine standards of the delivery suite. Following delivery, patients will be asked to complete a satisfaction questionnaire.
VAS pain score. | 12 month
  After giving consent, randomization will be carried out using sealed envelopes. After randomization women will be offered to withdraw consent. Women assigned to the study group will receive a sealed Laboraide™ package.
  Labor follow up will be documented regularly including outcome. The use of the DSD will not affect the regular management of labor according to the routine standards of the delivery suite. Following delivery, patients will be asked to complete a satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Yariv Yogev, professor, Principal Investigator — Director, Division of obstetrics and delivery
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel, Israel